CLINICAL TRIAL: NCT05097079
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Single-Treatment Efficacy and Safety Study of MYOBLOC® for the Treatment of Chronic Sialorrhea in Pediatric Subjects
Brief Title: Efficacy and Safety Study of MYOBLOC in the Treatment of Sialorrhea in Pediatric Subjects
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Company/sponsor business decision
Sponsor: Solstice Neurosciences, LLC, a subsidiary of MDD US Operations, LLC (Industry)
Responsible Party: Sponsor
Organization: Supernus Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SN-SIAL-302
Record Dates: First submitted 2021-10-18; First posted 2021-10-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Sialorrhea
MeSH Terms: conditions — Sialorrhea | interventions — rimabotulinumtoxinB

STUDY DESIGN:
Intervention Model Description: A Phase 3, multicenter, randomized, double-blind, placebo-controlled, single treatment study designed to assess the efficacy, safety, and tolerability of 2 dose levels of MYOBLOC compared to placebo for the treatment of chronic sialorrhea in pediatric subjects ages 3 to < 17 years.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MYOBLOC Low Dose (Experimental): MYOBLOC Low Dose will be administered as a single treatment via intraglandular injection (60 Units/kg)
  Interventions: Drug: MYOBLOC Low Dose
- MYOBLOC High Dose (Experimental): MYOBLOC High Dose will be administered as a single treatment via intraglandular injection (100 units/kg)
  Interventions: Drug: MYOBLOC High Dose
- Placebo (Placebo Comparator): Volume-matched placebo will be administered as a single treatment via intraglandular injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MYOBLOC Low Dose — Subjects assigned to the MYOBLOC Low Dose treatment group will be administered MYOBLOC (60 units/kg; maximum 1800 units) as a single treatment via intraglandular injection (5.0 units/kit per submandibular gland [maximum 150 units] and 25.0 units/kg per parotid gland [maximum 750 units])
  Other Names: rimabotulinumtoxinB
  Arms: MYOBLOC Low Dose
Drug: MYOBLOC High Dose — Subjects assigned to the MYOBLOC High Dose treatment group will be administered MYOBLOC (100 units/kg; maximum 3000 units) as a single treatment via intraglandular injection (25.0 units/kit per submandibular gland [maximum 300 units] and 40.0 units/kg per parotid gland [maximum 1200 units])
  Other Names: rimabotulinumtoxinB
  Arms: MYOBLOC High Dose
Drug: Placebo — Subjects assigned to the Placebo treatment group will be administered volume-matched placebo (1:1)
  Other Names: PBO
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of MYOBLOC for the treatment of chronic sialorrhea in pediatric subjects.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, single treatment study designed to assess the efficacy, safety, and tolerability of 2 dose levels of MYOBLOC vs placebo for the treatment of chronic sialorrhea in pediatric subjects ages 3 to < 17 years. Eligible subjects will be randomized 1:1:1 to receive single treatment of the low dose of MYOBLOC (60 Units/kg), the high dose of MYOBLOC (100 Units/kg), or volume-matched placebo via intraglandular injection.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject's parent or legally authorized representative(s) (LAR)/guardian(s) in accordance with local laws and Institutional Review Board (IRB)/Independent Ethics Committee (IEC) requirements.
2. Written minor assent obtained from the subject, as applicable and in accordance with local laws and IRB/IEC requirements.
3. Male or female ages 3 to < 17 years at the time of signing informed consent (and assent, if applicable) at Screening.
4. Minimum weight of 10 kg at Screening and Baseline (prior to randomization).
5. Chronic sialorrhea due to a neurological disorder (e.g., cerebral palsy (CP), or traumatic brain injury (TBI)) for at least 3 months prior to Screening.
6. A mTDS score ≥ 5 at Screening and Baseline (prior to randomization).
7. A minimum USFR of 0.2 g/min at Screening and Baseline (prior to randomization).
8. Females of childbearing potential (FOCP) must be either sexually inactive (abstinent) or, if sexually active, must agree to use/practice one of the following acceptable methods of contraception beginning during screening period prior to baseline (randomization, injection), for the duration of the study, and 2 months after study completion:

   1. simultaneous use of male condom and intra-uterine contraceptive device placed during screening period prior to baseline (randomization, injection)
   2. barrier method: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository;
   3. established use of oral, injected or implanted hormonal methods of contraception;
   4. surgically sterile male partner (e.g., vasectomized partner is sole partner). With approval by the Investigator, subjects' parents or legal guardians may select abstinence as a form of birth control if deemed more appropriate. For the purposes of this study, all females are considered to be of childbearing potential unless they are confirmed by the Investigator to be premenarchal, biologically sterile, or surgically sterile (e.g., hysterectomy with bilateral oophorectomy, tubal ligation).
9. Subject and the subject's parent/LAR are willing and able to comply with scheduled visits, treatment plan, laboratory tests, home monitoring, and other study procedures.

Exclusion Criteria:

1. FOCP subjects who are pregnant, lactating/breastfeeding and/or sexually active and not agreeing to use one of the acceptable birth control methods throughout the study.
2. History of drug or alcohol abuse within 6 months before Screening.
3. Treatment with an investigational drug, device, or biological agent within 30 days before Screening or while participating in this study.
4. Major surgery (requiring general anesthesia) within 3 months before screening, or any anticipated or scheduled surgery during the study period (with or without general anesthesia).
5. Aspiration pneumonia within 6 months before Screening.
6. History of moderate dysphagia or severe dysphagia (defined as an inability to swallow liquids, solids or both without choking or medical intervention) within 6 months before screening. Subjects who require gastrostomy tube feeding are not excluded provided tube placement was at least 30 days prior to Baseline (Day 1; injection).
7. Requires general anesthesia for study drug administration.
8. Prior botulinum toxin type A (BoNT/A) or BoNT/B treatment for sialorrhea or cervical dystonia within 20 weeks before screening. Prior BoNT/A or BoNT/B treatment in other anatomical locations is not exclusionary, but must have occurred at least 12 weeks prior to screening. Prior toxin exposure must have been well tolerated and without any significant long-term side effects in cases of repeated prior exposure.
9. Subjects must not receive nor have any plans to receive any other form of botulinum toxin treatment, other than the study drug (MYOBLOC), from the time that the informed consent is obtained until participation in the study is complete.
10. History of lack of response to MYOBLOC.
11. Any previous known or suspected hypersensitivity to botulinum toxins type A (BoNT/A) or B (BoNT/B) or to any of the MYOBLOC solution components.
12. Oxygen saturation < 95% on room air at Screening and Baseline (prior to randomization).
13. Subjects taking medications with anticholinergic/antihistamine properties who have not been on a stable dose and regimen for at least 2 weeks before Day 1. The same dose and dosing regimen must be maintained through the Week 4 study visit.
14. Diagnosed with Obstructive Sleep Apnea which requires nightly Continuous Positive Airway Pressure (CPAP) or Bi-level Positive Airway Pressure (BiPAP) therapy, such that subject has been receiving nightly therapy for at least 30 days.
15. Current or recent treatment (exposure within 5 half-lives of screening) or treatment at any time during the study with aminoglycoside antibiotics, curare-like agents, other agents that interfere with neuromuscular function, or dopamine receptor blocking agents (e.g., clozapine).
16. Current treatment or treatment at any time during the study with Coumadin® (warfarin) or similar anti-coagulant medications. Anti-platelet medications are not specifically exclusionary.
17. Prior surgery or irradiation in the head and neck to control sialorrhea (including salivary gland surgery or salivary gland irradiation) within 1 year before screening or planned during the study.
18. Extremely poor dental and/or oral condition, including infection at injection site(s) that might preclude safe study participation according to the judgment of the Investigator.
19. Has one or more screening clinical laboratory test values outside the reference range that, in the opinion of the Investigator, are clinical significant, or any of the following:

    1. Serum creatinine >1.5 times the upper limit of normal (ULN);
    2. Serum total bilirubin >1.5 times ULN;
    3. Serum alanine aminotransferase or aspartate aminotransferase >2 times ULN.
20. Has any of the following cardiac findings at Screening:

    1. Abnormal ECG that is, in the Investigator's opinion/evaluation, clinically significant;
    2. PR interval > 150 msec (2-5 years old); > 170 msec (6-11 years old); or > 180 msec (12-17 years old)
    3. QRS interval > 80 msec (2-5 years old); or > 90 msec (6-17 years old)
    4. QTcF interval >450 msec (for males), or >470 msec (for females) (QT corrected using Fridericia's method);
    5. Second-or third-degree atrioventricular block;
    6. Any rhythm, other than sinus rhythm, that is interpreted or assessed by the Investigator to be clinically significant.
21. Has received COVID-19 vaccine (single or 2nd dose) in the last 30 days prior to Screening.
22. Chronic or current use of inhaled corticosteroids, short acting beta-agonists or any other medication to manage asthma or other lung conditions such as emphysema.
23. Any other medical illness, condition, or clinical finding, including clinically significant abnormal laboratory values that in the opinion of the Investigator and/or the Sponsor, would put the subject at undue risk.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in the Unstimulated Saliva Flow Rate (USFR) at Week 4 post-injection. | Baseline and Week 4
  At each study visit, the subject's saliva is collected for at least 3 minutes and weighed (grams). The Unstimulated Saliva Flow Rate (USFR; grams/minute) for each visit is calculated for by dividing the 'total grams of saliva collected during the collection period' by the 'total minutes of the collection period. The USFR at Week 4 post-injection visit subtracted from the USFR at Baseline visit (prior to injection) yields the change from baseline USFR. A change from baseline USFR <0 grams/minutes represents a better outcome.
The Clinical Global Impression of Change (CGI-C) score at Week 4 post-injection. | Week 4
  The Clinical Global Impression of Change (CGI-C) scale is a single item clinician assessment of how much the subject's condition (sialorrhea) has improved, worsened or has not changed relative to subject's state at baseline prior to treatment (injection). The CGI-C is rated on a 7-point scale from 1 to 7, where 1 = "Very much improved", 2 = "Much improved", 3 = "Minimally improved", 4 = "No change", 5 = "Minimally worse", 6 = "Much worse", and 7 = "Very much worse". A CGI-C score <4 represents a better outcome.

SECONDARY OUTCOMES:
The Parent/Guardian Global Impression of Change (PGI-C) score at Week 4 post-injection. | Week 4
  The Parent/Guardian Global Impression of Change (PGI-C) scale is a single item parent/guardian assessment of how much the subject's condition (sialorrhea) has improved, worsened or has not changed relative to subject's state at baseline prior to treatment (injection). The PGI-C is rated on a 7-point scale from 1 to 7, where 1 = "Very much improved", 2 = "Much improved", 3 = "Minimally improved", 4 = "No change", 5 = "Minimally worse", 6 = "Much worse", and 7 = "Very much worse". A PGI-C score <4 represents a better outcome
The change from baseline in the Unstimulated Saliva Flow Rate (USFR) at Weeks 2, 8 and 13 post-injection. | Baseline and Weeks 2, 8 and 13
  At each study visit, the subject's saliva is collected for at least 3 minutes and weighed (grams). The Unstimulated Saliva Flow Rate (USFR; grams/minute) for each visit is calculated for by dividing the 'total grams of saliva collected during the collection period' by the 'total minutes of the collection period'. The USFR at the post-injection visit subtracted from the USFR at Baseline visit (prior to injection) yields the change from baseline USFR. A change from baseline USFR <0 grams/minutes represents a better outcome.
The Clinical Global Impression of Change (CGI-C) score at Weeks 2, 8, and 13 post-injection. | Weeks 2, 8 and 13
  The Clinical Global Impression of Change (CGI-C) scale is a single item clinician assessment of how much the subject's the subject's condition (sialorrhea) has improved, worsened or has not changed relative to subject's state at baseline prior to treatment (injection). The CGI-C is rated on a 7-point scale from 1 to 7, where 1 = "Very much improved", 2 = "Much improved", 3 = "Minimally improved", 4 = "No change", 5 = "Minimally worse", 6 = "Much worse", and 7 = "Very much worse". A CGI-C score <4 represents a better outcome.
The Parent/Guardian Global Impression of Change (PGI-C) score at Week 2, 8, and 13 post-injection. | Weeks 2, 8, and 13
  The Parent/Guardian Global Impression of Change (PGI-C) scale is a single item parent/guardian assessment of how much the subject's condition (sialorrhea) has improved, worsened or has not changed relative to subject's state at baseline prior to treatment (injection). The PGI-C is rated on a 7-point scale from 1 to 7, where 1 = "Very much improved", 2 = "Much improved", 3 = "Minimally improved", 4 = "No change", 5 = "Minimally worse", 6 = "Much worse", and 7 = "Very much worse". A PGI-C score <4 represents a better outcome.
The change from baseline in the Modified Teacher's Drooling Scale (mTDS) score at Week4 post injection. | Baseline and Week 4
  The Modified Teacher's Drooling Scale (mTDS) is a single-item scale used to assess subject's drooling severity and frequency. It is rated by the parent/guardian on a 9-point scale (1-9); where 1 = "Dry: never drools"; 2 = "Mild: only the lips are wet, occasionally"; 3 = "Mild: only the lips are wet, frequently"; 4 = "Moderate: wet on the lips and chin, occasionally"; 5 = "Moderate: wet on the lips and chin, frequently"; 6 = "Severe: drools to the extent that clothing becomes damp, occasionally"; 7 = "Severe: drools to the extent that clothing becomes damp, frequently"; 8 = "Profuse: clothing, hands, tray, and objects become wet, occasionally"; 9 = "Profuse: clothing, hands, tray, and objects become wet, frequently". The mTDS score at Week 4 Post injection subtracted from the mTDS score at Baseline yields the change from baseline mTDS score. A change from baseline mTDS score <0 represents a better outcome.
The change from baseline in the Drooling Impact Scale (DIS) score at Week 4 post-injection. | Baseline and Week 4
  The Drooling Impact Scale (DIS) is a 10-item questionnaire used to assess the frequency, severity, and impact of subject's drooling. Each item is rated by the parent/guardian on a 10-point end-anchor semantic differential scale (1 to 10; where 1 = "best outcome" to 10 = "worst outcome"). The sum of all 10 items yields a total score (ranging from 10-100). The DIS total score at Week 4 Post injection subtracted from the DIS total score at Baseline yields the change from baseline DIS total score. A change from baseline DIS score <0 represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rubin, MD, Study Director — Supernus Pharmaceuticals